CLINICAL TRIAL: NCT02961712
Title: Immunotherapy of Natural Killer in HTLV-1 Associated Myelopathy
Brief Title: Immunotherapy of Natural Killer(NK) Cells in Human T Lymphotropic Virus Type 1(HTLV-1) Associated Myelopathy(HAM)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Fujian Medical University (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK-HAM
Record Dates: First submitted 2016-11-03; First posted 2016-11-11 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2016-11

CONDITIONS: HAM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cell therapy (Experimental): NK cells and amniotic epithelial cells
  Interventions: Biological: NK cells; Biological: amniotic epithelial cells

INTERVENTIONS:
Biological: NK cells — single intravenous injection of NK cells (0.9~1*10^9)
Biological: amniotic epithelial cells — single intrathecal injection of amniotic epithelial cells

SUMMARY:
HTLV-1 Associated Myelopathy is a chronic disease of the spinal cord, caused by a virus called human T lymphotropic virus type 1（HTLV-1）. Natural Killer cells provide rapid responses to viral-infected cells, acting at around 3 days after infection, and respond to tumor formation. In this trial, the investigators aim to study the therapeutic safety and the effect on HTLV-1 virus. This in turn will improve the knowledge and understanding of the disease and should lead to better therapy.

DETAILED DESCRIPTION:
HAM is a chronic disease of the spinal cord, caused by a virus called HTLV-I. Natural Killer cells provide rapid responses to viral-infected cells, acting at around 3 days after infection, and respond to tumor formation. In this trial, the investigators aim to study the therapeutic safety and the effect on HTLV-1 virus. This in turn will improve the knowledge and understanding of the disease and should lead to better therapy.

In a single-center, one year open-label trial, 5 HAM patients will be treated with single intravenous injection of NK cells (0.9~1*10^9). Then, the the clinical effect was evaluated by dynamic analysis of Osame's Motor Disability Score and other related physiological indices, such as HTLV-1 antibody titer in blood and cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HTLV-1 associated myelopathy

Exclusion Criteria:

* HIV infection
* Hepatitis B & C viral infections
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
change of Osame's Motor Disability Score | 1 year
  The score were defined as follows: 0, no disability; 1, walking slow; 2, a little trouble when walking; 3, unable to run; 4, needs guardrail while going up the stairs; 5, needs one hand support while walking; 6, needs two hands support while walking (> 10 m); and 7, needs two hands support while walking (< 10 m); 8, needs two hands support while walking (< 5 m); 9, unable to walk but can crawl; 10, unable to crawl but can move; 11, unable to move but can roll over on the bed; 12 unable to roll over; 13, unable to flex toes

SECONDARY OUTCOMES:
HTLV-1 antibody titer in serum | 1 year
HTLV-1 antibody titer in cerebrospinal fluid | 1 year
HTLV-1 proviral load in blood | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhi Gao, Dr., Principal Investigator — The Second Affiliated Hospital of Fujian Medical University
Locations (1):
- The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided